CLINICAL TRIAL: NCT03391076
Title: The Clinical Value of FilmArray Rapid Viral Testing in Acute Hospitalized Lower Respiratory Infection Patients: A Randomized Controlled Study
Brief Title: The Clinical Value of FA in AHLRI Patients
Acronym: FALRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bin Cao (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor-Investigator, Bin Cao, Head of Respiratory Department, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20170909
Record Dates: First submitted 2017-12-07; First posted 2018-01-05 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Lower Respiratory Tract Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- FilmArray group (Experimental): Patients in this group will use FilmArray Respiratory Panel to test potential viral pathogens.
  Interventions: Diagnostic Test: FilmArray Respiratory Panel
- Routine test group (No Intervention): Patients in this group will use clinical routine methods to test potential viral pathogens.

INTERVENTIONS:
Diagnostic Test: FilmArray Respiratory Panel — An Multi-PCR method which can detect 20 pathogens in 45 minutes.
  Arms: FilmArray group

SUMMARY:
LRTI (Lower respiratory tract infection) is a severe disease in China. The fast and accurate diagnosis of pathogens, bacteria or viruses that cause the infection is critical for the therapy. In this study, investigators assume that the use of FilmArray Respiratory Panel will provide more rapid and comprehensive evidences to physicians to diagnose LRTI which is caused by viruses or atypical pathogens and then reduce the length of antibiotics use by 0.5-1.0 days as well as other hospital resources (length of hospital/ICU stay, take-away oral antibiotics, etc.). Secondly, investigators assume that in LRTI patients with viral infection and a low serum PCT level, fewer length of antibiotics use can be expected. Thirdly, the use of FilmArray Respiratory Panel will provide clearer epidemiology data of virus and atypical pathogens in hospitalized LRTI patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults age >= 18 years old
* Community acquired Pneumonia, acute exacerbation of chronic obstructive pulmonary disease [AECOPD], acute exacerbation of bronchiectasis.
* Hospitalization required
* Informed Consent Form signed

Exclusion Criteria:

* Age < 18 years old
* Hospital acquired Pneumonia
* Patients with lung tuberculosis
* Pregnant women
* Patients with immunodeficiency
* Any conditions which may increase PCT levels
* Informed Consent Form not signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-10-23 (Estimated)

PRIMARY OUTCOMES:
The length (days) of antibiotics therapy in hospital between two groups. | From in-hospital to discharge or death, whichever came first, assessed up to 12 months
  The duration of antibiotics used is defined as days of intravenous antibiotic therapy in which any doses of antibiotics are administered.

SECONDARY OUTCOMES:
Antibiotics therapy cost | From in-hospital to discharge or death, whichever came first, assessed up to 12 months
Length of hospital stay (LOS) and/or ICU stay | From in-hospital to discharge or death, whichever came first, assessed up to 12 months
The correlation between the initial serum PCT level and clinical outcomes/mortality | From in-hospital to discharge or death, whichever came first, assessed up to 12 months
The detection rate of viruses and atypical pathogens by FilmArray in LRTI patients | From in-hospital to discharge or death, whichever came first, assessed up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chian Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shengchen D, Gu X, Fan G, Sun R, Wang Y, Yu D, Li H, Zhou F, Xiong Z, Lu B, Zhu G, Cao B. Evaluation of a molecular point-of-care testing for viral and atypical pathogens on intravenous antibiotic duration in hospitalized adults with lower respiratory tract infection: a randomized clinical trial. Clin Microbiol Infect. 2019 Nov;25(11):1415-1421. doi: 10.1016/j.cmi.2019.06.012. Epub 2019 Jun 20. PMID 31229593